CLINICAL TRIAL: NCT00885599
Title: A Randomized Multi-treatment/Controlled Double-blinded Study to Evaluate the Efficacy of a Naturally-derived Mouthrinse in the Treatment of Gingival Inflammation.
Brief Title: Efficacy of a Naturally-derived Mouthrinse for Gingival Inflammation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Menachem Oberbaum, Director, Center for Integrative Complementary Medicine, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gingival-ST2
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Gingivitis
Keywords: gingivitis; natural remedy; inflammation; C-reactive protein; mouthwash
MeSH Terms: conditions — Gingivitis; Inflammation | interventions — Benzocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PERIORINSE (Experimental): naturopathic remedy
  Interventions: Drug: Herbal API
- CPC (Active Comparator): Cepacol, standard anti-bacterial mouthwash
  Interventions: Drug: Cepacol
- Listerine (Active Comparator): standard anti-bacterial mouthwash
  Interventions: Drug: Listerine Antiseptic Mouth Rinse
- placebo (Placebo Comparator): colored water
  Interventions: Drug: placebo mouthwash

INTERVENTIONS:
Drug: Herbal API — mouthwash;rinse full strength for 30 seconds with 20 ml (2/3 fl. Ounce or 4 teaspoonfuls) morning and night.
  Arms: PERIORINSE
Drug: Cepacol — mouthwash;rinse full strength for 30 seconds with 20 ml (2/3 fl. Ounce or 4 teaspoonfuls) morning and night.
  Arms: CPC
Drug: Listerine Antiseptic Mouth Rinse — mouthwash;rinse full strength for 30 seconds with 20 ml (2/3 fl. Ounce or 4 teaspoonfuls) morning and night.
  Arms: Listerine
Drug: placebo mouthwash — colored water mouthwash;rinse full strength for 30 seconds with 20 ml (2/3 fl. Ounce or 4 teaspoonfuls) morning and night.
  Arms: placebo

SUMMARY:
Gingivitis, defined as inflammation of the gingival tissues, has long been associated with bacterial accumulation [plaque] on the tooth surface adjacent to the gingiva, causing an inflammatory reaction. Experimental gingivitis in health adults can be induced by abstension from brushing teeth for 9 to 21 days, and can test the effects of numerous chemotherapeutic agents, rinses and toothpastes. Effective prevention of plaque accumulation can prevent destructive forms of periodontal disease.

A recent link has been established between localized gingival inflammation and systemic inflammation and a number of disease processes. Periodontal disease may lead to elevated C-reactive protein [CRP], considered a potential risk factor for cardiovascular disease and stroke. It has been shown that reducing gingival inflammation is accompanied with a significant decrease in serum CRP levels.

Naturopathic remedies for treating oral disease have been well documented in the medical and dental literature since early civilization, and have become more and more popular in recent years. We propose to study one such remedy, PERIORINSE. This remedy consists of a number of herbs, and has been shown to exhibit antibacterial and anti-inflammatory effects. Specifically, it has been shown to block the proteolytic effects seen in gingival inflammation . This study will evaluate the efficacy of this formulation, using currently accepted clinical testing protocols.

A Random sample of 100 healthy volunteers who fulfill all inclusion criteria and no exclusion criteria, will be included in the study. Patients will randomly selected to one of 4 treatment groups: PERIORINSE (n=25), CPC (Cepacol) mouthwash (25 patients), Listerine mouthwash (n=25), and placebo (colored water) mouthrinse. Patients will be examined at baseline, and Gingival Index taken for all teeth. A blood specimen will be taken to measure CRP levels as well. Patients will be given a full dental prophylaxis which includes scaling and tooth polishing, and given rinsing instructions and reminded to cease all other oral hygiene methods including brushing, flossing, and rinsing with any other rinse for a period of 14 days. On day 14, patients will be re-examined and Gingival Index taken for all teeth. Patients will be given a full dental prophylaxis which includes scaling and tooth polishing and required to reinstitute their original oral hygiene regimen. CRP levels will be measured again, as well.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-75.
* Clinical diagnosis of Gingivitis as measured by the Gingival index ≤ 0.5
* Healthy volunteer willing to cease all oral hygiene methods except for the mouthrinse for a period of three weeks.
* Have at least 24 teeth in their mouth

Exclusion Criteria:

* Pregnant or planning to become pregnant during the study period.
* Periodontal pockets greater than 5mm in 3 or more areas.
* History of periodontal treatment within the last month.
* Antibiotic treatment within the last month
* Use of any antimicrobial mouthrinse within the last month.
* Participation in another trial within one month prior to the study.
* Inability to comply with the trial protocol by not rinsing with mouthrinse 20% of time.
* Inability to comply, brushing the teeth or using another mouthrinse during the study period.
* Systemic Disease.
* On antibiotic or anti-inflammatory medication
* Cigarette-smoking

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Difference in the Gingival Index scores between the start and the end of the study | 14 days

SECONDARY OUTCOMES:
The difference in C-Reactive protein levels between the start and the end of the study. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel